CLINICAL TRIAL: NCT03777176
Title: A Two-Period, Open-label Trial Evaluating the Efficacy and Safety of Dasiglucagon for the Treatment of Children With Congenital Hyperinsulinism
Brief Title: A Two-Period Open-label Trial Evaluating Efficacy and Safety of Dasiglucagon in Children With Congenital Hyperinsulinism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZP4207-17109
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Congenital Hyperinsulinism
MeSH Terms: conditions — Congenital Hyperinsulinism | interventions — dasiglucagon; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care + dasiglucagon (Experimental): 4 weeks (Treatment Period 1) + 4 weeks (Treatment Period 2) of dasiglucagon treatment as an SC infusion starting at 10 µg/hr on top of standard of care
  Interventions: Drug: Dasiglucagon; Other: Standard of Care
- Standard of Care Only (Other): 4 weeks (Treatment Period 1) of standard of care only + 4 weeks (Treatment Period 2) of dasiglucagon treatment as an SC infusion starting at 10 µg/hr on top of standard of care
  Interventions: Drug: Dasiglucagon; Other: Standard of Care

INTERVENTIONS:
Drug: Dasiglucagon — Glucagon analog
  Other Names: ZP4207
Other: Standard of Care — Standard of care according to site and/or country

SUMMARY:
The objective of the trial is to evaluate the efficacy and safety of dasiglucagon administered as a subcutaneous (SC) infusion in reducing hypoglycemia in children with CHI.

ELIGIBILITY:
Inclusion Criteria:

* Established and documented diagnosis of CHI based on standard of care
* Experiencing ≥3 events of hypoglycemia per week (plasma glucose [PG] <70 mg/dL [<3.9 mmol/L]) according to the investigator's evaluation
* Previously undergone near-total pancreatectomy or being treated with a non-surgical approach, having been evaluated as not eligible for pancreatic surgery
* If somatostatin analogues or sirolimus are used, the therapy should be well established as judged by the investigator, especially when considering their biological half-life

Exclusion Criteria:

* Previous administration of dasiglucagon
* Known or suspected allergy to the trial drug or related products
* Previous participation (randomization) in this trial
* Circulatory instability requiring supportive medication or presence of pheochromocytoma
* Requires exogenous insulin
* Body weight of <4 kg (8.8 lbs.)
* Documented HbA1c ≥7% subsequent to near-total pancreatectomy and within 6 months prior to screening
* Known or suspected presence of significant central nervous system disease/injury such that in the investigator's opinion will affect trial participation
* Use of systemic corticosteroids, e.g., hydrocortisone >20 mg/m2 body surface area or equivalent in the 5 days before screening
* Use of anti-inflammatory biological agents, or other immune modulating agents in the 3 months prior to screening
* Any clinically significant abnormality identified on echocardiogram that in the opinion of the investigator would affect the patient's ability to participate in the trial
* Any recognized clotting or bleeding disorders
* Has participated in an interventional clinical trial (investigational or marketed product) within 3 months of screening or 5 half-lives of the drug under investigation (whichever comes first), or plans to participate in another clinical trial.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Teglman Schioeler, Study Director — Zealand Pharma
Locations (10):
- United States (3):
  - Children's Hospital of Colorado, Aurora, Colorado
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Germany (2):
  - University Hospital Düsseldorf, Department of Pediatrics, Düsseldorf
  - Otto von Guericke University Magdeburg, Department of Pediatrics, Magdeburg
- Hadassah Medical Center, Jerusalem, Israel
- United Kingdom (4):
  - NHS Greater Glasgow and Clyde, Glasgow
  - Alder Hey Children'sHospital NHS Foundation Trust, Liverpool
  - Great Osmond Street Hospital for Children NHS Foundation Trust, London
  - Central Manchester University Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care + Dasiglucagon (Treatment Period 1): 4 weeks (Treatment Period 1) of dasiglucagon treatment as an SC infusion starting at 10 µg/hr on top of standard of care
  Dasiglucagon: Glucagon analog
  Standard of care: Standard of care according to site and/or country
- Standard of Care Only (Treatment Period 1): 4 weeks (Treatment Period 1) of standard of care only
  Standard of care: Standard of care according to site and/or country
- Standard of Care + Dasiglucagon (Treatment Period 2): 4 weeks (Treatment Period 2) of dasiglucagon treatment as an SC infusion starting at 10 µg/hr on top of standard of care
  Dasiglucagon: Glucagon analog
  Standard of care: Standard of care according to site and/or country
Period: Treatment Period 1
Arm/Group | Standard of Care + Dasiglucagon (Treatment Period 1) | Standard of Care Only (Treatment Period 1) | Standard of Care + Dasiglucagon (Treatment Period 2)
Started | 16 | 16 | 0 (This arm was not applicable to Treatment Period 1.)
Completed | 16 | 16 | 0
Not Completed | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Standard of Care + Dasiglucagon (Treatment Period 1) | Standard of Care Only (Treatment Period 1) | Standard of Care + Dasiglucagon (Treatment Period 2)
Started | 0 (This arm was not applicable to Treatment Period 2.) | 0 (This arm was not applicable to Treatment Period 2.) | 32
Completed Study But Discontinued Treatment Due to an AE | 0 | 0 | 1
Completed | 0 | 0 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Only: 4 weeks (Treatment Period 1) of standard of care + 4 weeks (Treatment Period 2) of dasiglucagon treatment as an SC infusion starting at 10 µg/hr on top of standard of care
  Dasiglucagon: Glucagon analog
  Standard of care: Standard of care according to site and/or country
- Total: Total of all reporting groups
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.55 (2.592) | 5.00 (2.892) | 4.27 (2.800)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 12 | 16 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14
  United Kingdom | 6 | 3 | 9
  Israel | 0 | 3 | 3
  Germany | 3 | 3 | 6
Gastrostomy/nasogastric tube [Count of Participants; unit: Participants]
  Gastrostomy | 9 | 12 | 21
  Nasogastric tube | 2 | 1 | 3
  None | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemia Episode Rate
Description: Hypoglycemia episode rate, defined as average weekly number of hypoglycemic episodes (PG <70 mg/dL [3.9 mmol/L]) during Weeks 2-4 as detected by self-monitored plasma glucose (SMPG). The Week 2-4 value is the average weekly number of hypoglycemic episodes across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the average weekly number of hypoglycemic episodes during the 2-week baseline period.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 16 | 16
episodes per week
  Weekly number of episodes in Weeks 2-4 | 5.29 (5.256) | 5.85 (2.767)
  Change from Baseline | -3.05 (4.343) | -3.15 (4.753)
Statistical Analysis 1: Comparison: Standard of Care + Dasiglucagon vs Standard of Care Only; The primary analysis was performed as a negative binominal regression analysis on the difference of the SMPG-detected hypoglycemia episode rate between treatment groups over the Weeks 2-4; Test type: Superiority — The negative binomial regression used region and treatment group as fixed effects, and Baseline hypoglycemic rate as covariate and number of hypoglycemic events during Weeks 2-4 as dependent variable; p = 0.5028, Negative binomial regression; Event rate ratio = 0.85, 95% CI 2-sided [0.54 to 1.36]

2. Secondary Outcome: Increase in Fasting Tolerance
Description: Increase in fasting tolerance (time from beginning of meal to the beginning of the first continuous 15-minute continuous glucose monitoring reading <70 mg/dL [3.9 mmol/L]), or the time the test ended if a continuous 15-minute CGM reading <70 mg/dL was not reached. The change from Baseline to the End of Treatment Period 1 (Week 4) is also provided. The Baseline value is the value recorded at the Screening visit.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: There were 2 missing values at the end of Treatment Period 1 in the dasiglucagon + standard of care group.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 14 | 16
hours
  End of Treatment Period 1 | 6.13 (5.335) | 4.22 (4.222)
  Change from Baseline | 1.20 (5.908) | 1.27 (3.836)
Statistical Analysis 1: Comparison: Standard of Care + Dasiglucagon vs Standard of Care Only; Test type: Superiority; p = 0.6433, ANCOVA — The P value should be interpreted with caution given the procedural issues (hypoglycemia at the beginning of the test, test meals not being the same, and some children only having 1 test) which affected the preplanned statistical evaluation; Mean Difference (Net) = 0.84, 95% CI 2-sided [-2.71 to 4.39]

3. Secondary Outcome: Percent Time in Range 70-180 mg/dL
Description: Percent time in range 70-180 mg/dL (3.9-10.0 mmol/L) during Weeks 2-4 as measured by continuous glucose monitoring. The Week 2-4 value is the average weekly percent time in range 70-180 mg/dL across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value was calculated as the average percent time in range during the 14 days before randomization.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: There was 1 missing value at Baseline for the dasiglucagon + standard of care group.
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 16 | 16
percent time
  Week 2-4 | 75.10 (11.821) | 72.65 (7.313)
  Change from Baseline: number analyzed (Participants) | 15 | 16
  Change from Baseline | -0.97 (11.837) | 2.44 (9.584)
Statistical Analysis 1: Comparison: Standard of Care + Dasiglucagon vs Standard of Care Only; Test type: Superiority; p = 0.9653, ANCOVA — There was 1 missing value at Baseline for the dasiglucagon + standard of care group; Mean Difference (Net) = 0.15, 95% CI 2-sided [-6.48 to 6.78]

4. Secondary Outcome: Clinically Significant Hypoglycemia Episode Rates
Description: Clinically significant hypoglycemia episode rates during Weeks 2-4, defined as average weekly number of clinically significant hypoglycemic episodes (PG <54 mg/dL [3.0 mmol/L]), as detected by SMPG. The Week 2-4 value is the average weekly clinically significant hypoglycemia episode rate across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the average weekly number of clinically significant hypoglycemic episodes during the 2-week baseline period.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 16 | 16
episodes per week
  Weekly number of episodes in Weeks 2-4 | 1.77 (1.857) | 1.90 (1.407)
  Change from Baseline | -0.51 (2.798) | -0.35 (1.446)
Statistical Analysis 1: Comparison: Standard of Care + Dasiglucagon vs Standard of Care Only; Test type: Superiority; p = 0.8114, Negative binominal regression; The negative binomial regression used region and treatment group as fixed effects, and Baseline hypoglycemic rate as covariate; Event rate ratio = 0.93, 95% CI 2-sided [0.49 to 1.74]

5. Secondary Outcome: Total Amount of Gastric Carbohydrates Administered to Treat Hypoglycemia
Description: Total amount of gastric carbohydrates administered via nasogastric tube or gastrostomy per week to treat hypoglycemia. The Week 2-4 value is the average weekly total amount of gastric carbohydrates across the last 3 weeks of treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the value recorded during the 2-week Baseline period.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: The total amount of gastric carbohydrates administered to treat hypoglycemia could be evaluated only in patients with gastrostomy or NG-tube at screening, and is summarized accordingly.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 11 | 13
grams
  Week 2-4 | 22.89 (31.415) | 37.66 (57.998)
  Change from Baseline | -33.66 (82.767) | -19.74 (64.082)

6. Secondary Outcome: Rate of Gastric Carbohydrates Administrations to Treat Hypoglycemia
Description: Rate of gastric carbohydrate administrations via nasogastric tube or gastrostomy per week to treat hypoglycemia, calculated as the number of times gastric carbohydrates were administered to treat hypoglycemia per week. The Week 2-4 value is the average weekly rate of gastric carbohydrate administrations across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the value recorded during the 2-week Baseline period.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of administrations per week
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 11 | 13
number of administrations per week
  Week 2-4 | 2.30 (3.433) | 2.18 (2.714)
  Change from Baseline | -0.29 (4.920) | -2.13 (3.825)

7. Secondary Outcome: Extent of Hypoglycemia
Description: Extent of hypoglycemia (area over the glucose curve [AOCglucose] below 70 mg/dL [3.9 mmol/L]) and below 54 mg/dL [3.0 mmol/L] as measured by continuous glucose monitoring. The extent of hypoglycemia was defined as the AOCglucose under the threshold divided by total duration in hours of CGM measurement. A reduction in this measure indicates a benefit. The Week 2-4 value is the average weekly extent of hypoglycemia below 70 mg/dL and below 54 mg/dL across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the value assessed during the 14 days before randomization.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: There was 1 missing value at Baseline for the dasiglucagon + standard of care group.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 16 | 16
mmol/L
  Week 2-4: Extent of Hypoglycemia Below 70 mg/dL (3.9 mmol/L) | 0.083 (0.0618) | 0.147 (0.0736)
  Change from Baseline in Extent of Hypoglycemia Below 70 mg/dL (3.9 mmol/L): number analyzed (Participants) | 15 | 16
  Change from Baseline in Extent of Hypoglycemia Below 70 mg/dL (3.9 mmol/L) | -0.062 (0.1003) | -0.019 (0.0959)
  Week 2-4: Extent of Hypoglycemia Below 54 mg/dL (3.0 mmol/L) | 0.015 (0.0117) | 0.025 (0.0132)
  Change from Baseline in Extent of Hypoglycemia Below 54 mg/dL (3.0 mmol/L): number analyzed (Participants) | 15 | 16
  Change from Baseline in Extent of Hypoglycemia Below 54 mg/dL (3.0 mmol/L) | -0.008 (0.0252) | -0.007 (0.0252)

8. Secondary Outcome: Amount of Nightly Gastric Carbohydrates Administered
Description: Amount of nightly (midnight to 6 am) gastric carbohydrates administered via nasogastric tube or gastrostomy per week. The change from Baseline is also provided for each week. The Baseline value is the value recorded during the 2-week Baseline period.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 11 | 13
grams
  Week 1 | 95.98 (153.272) | 33.43 (90.955)
  Change from Baseline at Week 1 | 41.64 (63.484) | 3.64 (27.29)
  Week 2 | 77.24 (147.065) | 39.25 (100.638)
  Change from Baseline at Week 2 | 22.90 (137.325) | 9.46 (40.853)
  Week 3 | 67.59 (141.062) | 30.31 (94.870)
  Change from Baseline at Week 3 | 13.24 (148.569) | 0.52 (25.022)
  Week 4 | 63.89 (127.849) | 34.62 (94.549)
  Change from Baseline at Week 4 | 9.55 (134.369) | 4.83 (25.689)

9. Secondary Outcome: Total Amount of Gastric Carbohydrates Administered
Description: Total amount of gastric carbohydrates administered (regardless of whether this was to treat hypoglycemia or not) via nasogastric tube or gastrostomy per week. The Week 2-4 value is the average amount of gastric carbohydrates administered via nasogastric tube or gastrostomy across the last 3 weeks of the treatment period. The change from baseline to Week 2-4 is also provided. The baseline value is the value recorded during the 2-week baseline period.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 11 | 13
grams
  Week 2-4 | 567.35 (453.373) | 775.96 (551.640)
  Change from Baseline | -146.56 (222.995) | 160.44 (438.735)

10. Secondary Outcome: Percent Time in Hypoglycemia
Description: Percent time in hypoglycemia (PG <70 mg/dL [3.9 mmol/L]) as measured by continuous glucose monitoring. The Week 2-4 value is the average weekly percent of time in hypoglycemia across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the value assessed during the 14 days before randomization.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: There was 1 missing value at Baseline for the dasiglucagon + standard of care group.
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 16 | 16
percent time
  Week 2-4 | 11.77 (9.248) | 20.22 (10.034)
  Change from Baseline: number analyzed (Participants) | 15 | 16
  Change from Baseline | -9.91 (10.119) | -1.95 (10.186)

11. Secondary Outcome: Rate of Hypoglycemic Episodes
Description: Rate of hypoglycemic episodes, defined as number of episodes with PG <70 mg/dL (3.9 mmol/L) for 15 minutes or more per week, as measured by continuous glucose monitoring. The Week 2-4 value is the average weekly number of hypoglycemic episodes across the last 3 weeks of the treatment period. The change from Baseline to Week 2-4 is also provided. The Baseline value is the average weekly number of hypoglycemic episodes during the 14 days before randomization.
Time Frame: Baseline, Week 2-4 (Treatment Period 1)
Population: There was 1 missing value at Baseline for the dasiglucagon + standard of care group.
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Standard of Care + Dasiglucagon | Standard of Care Only
Number analyzed (Participants) | 16 | 16
episodes per week
  Week 2-4 | 21.71 (14.179) | 36.88 (15.023)
  Change from Baseline: number analyzed (Participants) | 15 | 16
  Change from Baseline | -14.37 (21.184) | -6.28 (20.565)

12. Secondary Outcome: Percent Time in Hypoglycemia in Treatment Period 2
Description: Percent time in hypoglycemia (PG <70 mg/dL [3.9 mmol/L]) as measured by continuous glucose monitoring. The Week 6-8 value is the average weekly percent of time in hypoglycemia across the last 3 weeks of the treatment period. The change from Baseline to Week 6-8 is also provided. The Baseline value is the value assessed during the 14 days before randomization.
Time Frame: Baseline, Week 6-8 (Treatment Period 2)
Population: There was 1 participant with a missing value at Baseline.
Measure: Mean (Standard Deviation); unit: percent time
Arm/Group | Standard of Care + Dasiglucagon (Treatment Period 2)
Number analyzed (Participants) | 32
percent time
  Week 6-8 | 8.64 (6.011)
  Change from Baseline: number analyzed (Participants) | 31
  Change from Baseline | -13.27 (10.120)

13. Secondary Outcome: Rate of Gastric Carbohydrates Administrations to Treat Hypoglycemia in Treatment Period 2
Description: Rate of gastric carbohydrate administrations via nasogastric tube or gastrostomy per week to treat hypoglycemia, calculated as the number of times gastric carbohydrates were administered to treat hypoglycemia per week. The Week 6-8 value is the average weekly rate of gastric carbohydrate administrations across the last 3 weeks of the treatment period. The change from Baseline to Week 6-8 is also provided. The Baseline value is the value recorded during the 2-week Baseline period.
Time Frame: Baseline, Week 6-8 (Treatment Period 2)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of administrations per week
Arm/Group | Standard of Care + Dasiglucagon (Treatment Period 2)
Number analyzed (Participants) | 24
number of administrations per week
  Week 6-8 | 1.31 (2.254)
  Change from Baseline | -2.22 (4.990)

14. Secondary Outcome: Rate of Hypoglycemic Episodes in Treatment Period 2
Description: Hypoglycemia episode rate, defined as average weekly number of hypoglycemic episodes (PG <70 mg/dL [3.9 mmol/L]) as detected by SMPG. The Week 6-8 value is the average weekly number of hypoglycemic episodes across the last 3 weeks of the treatment period. The change from Baseline to Week 6-8 is also provided. The Baseline value is the average weekly number of hypoglycemic episodes during the 2-week baseline period.
Time Frame: Baseline, Week 6-8 (Treatment Period 2)
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Standard of Care + Dasiglucagon (Treatment Period 2)
Number analyzed (Participants) | 32
episodes per week
  Weekly number of episodes in Weeks 6-8 | 3.06 (2.730)
  Change from Baseline | -5.61 (4.096)

15. Secondary Outcome: Rate of Clinically Significant Hypoglycemia Episodes in Treatment Period 2
Description: Change from Baseline to Week 6-8 in the clinically significant (CS) hypoglycemia episode rate in treatment period 2, defined as the average weekly number of episodes <54 mg/dL (3.0 mmol/L), for 15 minutes or more, as measured by continuous glucose monitoring (CGM). The Week 6-8 value is the average weekly CS hypoglycemia episode rate across the last 3 weeks of the treatment period. The Baseline value is the average weekly number of CS hypoglycemic episodes during the 14 days before randomization.
Time Frame: Baseline, Week 6-8 (Treatment Period 2)
Population: There was 1 participant with a missing value at Baseline.
Measure: Mean (Standard Deviation); unit: episodes per week
Arm/Group | Standard of Care + Dasiglucagon (Treatment Period 2)
Number analyzed (Participants) | 32
episodes per week
  Week 6-8 | 7.78 (5.226)
  Change from Baseline: number analyzed (Participants) | 31
  Change from Baseline | -8.51 (9.941)

ADVERSE EVENTS:
Time Frame: Adverse event data were recorded from the time a signed and dated informed consent form was obtained until the end of the posttreatment follow-up period or inclusion in the ZP4207-17106 extension trial (up to 16 weeks, from Day -28 through Week 12).
Groups:
- Treatment Period 1: Standard of Care + Dasiglucagon: All participants treated with standard of care + dasiglucagon during Treatment Period 1 (Weeks 1 to 4)
  Dasiglucagon: Glucagon analog
  Standard of care: Standard of care according to site and/or country
- Treatment Period 1: Standard of Care Only: All participants treated with standard of care only during Treatment Period 1 (Weeks 1 to 4)
  Standard of Care: Standard of care according to site and/or country
- Treatment Period 2: Standard of Care + Dasiglucagon: All participants treated with standard of care + dasiglucagon during Treatment Period 2 (Weeks 5 to 8)
  Dasiglucagon: Glucagon analog
  Standard of care: Standard of care according to site and/or country
Arm/Group | Treatment Period 1: Standard of Care + Dasiglucagon | Treatment Period 1: Standard of Care Only | Treatment Period 2: Standard of Care + Dasiglucagon
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/32
Serious Adverse Events (participants affected / at risk) | 2/16 | 1/16 | 2/32
Other Adverse Events (participants affected / at risk) | 14/16 | 8/16 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1: Standard of Care + Dasiglucagon (N=16) | Treatment Period 1: Standard of Care Only (N=16) | Treatment Period 2: Standard of Care + Dasiglucagon (N=32)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vascular Device Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
H1N1 Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period 1: Standard of Care + Dasiglucagon (N=16) | Treatment Period 1: Standard of Care Only (N=16) | Treatment Period 2: Standard of Care + Dasiglucagon (N=32)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Localised Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Candida Nappy Rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eczema Infected (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Periorbital Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Necrolytic Migratory Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7) | 1 (1) | 2 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Post-Tussive Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Medical Device Site Irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter Site Haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1)
Developmental Delay (General disorders) | 0 (0) | 0 (0) | 1 (2)
Infusion Site Bruising (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Iron Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glycosylated Haemoglobin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Eye Movement Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (16)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stoma Site Hypergranulation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic Dilatation (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT03777176/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/76/NCT03777176/SAP_001.pdf